CLINICAL TRIAL: NCT04041479
Title: Efficacy of Biomarker-guided rTMS for Treatment Resistant Depression
Brief Title: Biomarker-guided rTMS for Treatment Resistant Depression
Acronym: BioTMS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-08023811; prev 1810019638; R01MH118388 (NIH)
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Human subjects in the proposed protocol will be randomized to receive a) biotype-guided rTMS to the left DLPFC or to the DMPFC; b) rTMS targeted to the opposite site; and c) standard-of-care left DLPFC rTMS. The dosage and method of delivery of rTMS are as follows: intermittent theta burst stimulation (iTBS) will be delivered at 120% of the resting motor threshold. It will be administered in triplet 50 Hz bursts, repeated at 5 Hz with a duty cycle of 2 s on and 8 s off, for a total of 600 pulses per session and a total duration of 3 min 9 s. Participants will receive screening and diagnostic interviews, phenotypic assessment (including demographic information, cognitive assessments, and behavioral functioning), structured clinical interviews, and magnetic resonance imaging (including structural and functional MRI).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Standard of Care (Active Comparator): FDA-cleared, standard-of-care iTBS repetitive Transcranial Magnetic Stimulation targeting the left dorsolateral prefrontal cortex (DLPFC), regardless of the depression subtype (biotype) determined by a magnetic resonance imaging (MRI) scan.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Targeted Side Arm (Experimental): iTBS rTMS targeting the area of the brain (DLPFC or dorsomedial prefrontal cortex DMPFC)) that we hypothesize will be most effective for that subject's biotype (confirmation arm).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Opposite Side Arm (Active Comparator): iTBS rTMS targeting the opposite site (DLPFC or DMPFC) than the one we hypothesize will be most effective for that subject's biotype (disconfirmation arm).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — iTBS rTMS targeting the DMPFC or left DLPFC
  Arms: Opposite Side Arm; Targeted Side Arm
Device: Repetitive Transcranial Magnetic Stimulation — iTBS rTMS targeting the left DLPFC
  Arms: Standard of Care

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is a treatment for depression. The investigators are continuing to learn how to optimize outcomes from rTMS treatment. The purpose of this research project is to use brain network connectivity patterns as measured by resting state functional magnetic resonance imaging (fMRI) to confirm a way to optimize the use of rTMS to treat depression. In addition, the study aims to gain a better understanding of how rTMS influences brain networks.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a leading cause of global disability, and approximately 30% of MDD patients are resistant to antidepressant pharmacotherapy. Repetitive transcranial magnetic stimulation (rTMS) of the left dorsolateral prefrontal cortex (DLPFC) is an FDA-cleared intervention with proven efficacy in treatment-resistant depression, but only 30-40% of these patients achieve remission after a single course. Other studies have shown that rTMS targeting the dorsomedial prefrontal cortex (DMPFC) is comparably effective, but biomarkers for informing target site selection do not exist. Diagnostic heterogeneity has been an obstacle to biomarker discovery efforts. Recently, we developed and validated an approach to diagnose four novel MDD subtypes or "biotypes' defined by resting state functional connectivity (RSFC) patterns and predicting differing antidepressant responses at the individual level to rTMS. This pivotal trial will test a novel, biotype-guided treatment selection strategy motivated by the hypothesis that an individual patient's likelihood of responding to left DLFPC vs.DMPFC rTMS is determined in part by individual differences in 1) the degree to which their symptoms are driven by dysfunction in specific cerebral network targets comprising Valence Systems; and 2) the degree to which dysfunction in those targets can be modulated by stimulating the left DLPFC or DMPFC. Subjects (N=348; 174 from this site) will be randomized to receive a) biotype-guided rTMS targeting the DMPFC or left DLPFC; b) to a disconfirmation arm receiving rTMS targeting the opposite site; and c) to a third arm receiving FDA-cleared, standard-of-care rTMS targeting the left DLFPC, regardless of biotype. The dosage and method of delivery of rTMS for all arms are as follows: intermittent theta burst stimulation (iTBS) will be delivered at 120% of the resting motor threshold. It will be administered in triplet 50 Hz bursts, repeated at 5 Hz with a duty cycle of 2 s on and 8 s off, for a total of 600 pulses per session and a total duration of 3 min 9 s. All patients will be assessed before and after treatment on a battery of fMRI, behavioral, and clinical assessments. The primary goal is to confirm the efficacy of a novel RSFC biomarker-guided approach to differential treatment selection in treatment resistant depression.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 to 65 years
* Major Depressive Disorder (by M.I.N.I., Diagnostic Statistical Manual V (DSM-V criteria)); Verification by evaluation by licensed study psychiatrist or psychologist
* At least moderately severe depression (17-item Hamilton Depression Rating Scale greater than or equal to 18)
* Failure to respond in the current episode to at least 1 antidepressant medication at an adequate dose and duration as measured by a modified Antidepressant Treatment History Form. The Maudsley Staging Method will also be used to quantify treatment resistance.
* Any and all medication intended to treat depression or reduce symptoms of depression must be discontinued or maintained at the same daily dose for ≥ 4 weeks prior to enrollment and for the duration of the study
* Capacity to consent
* Written consent to allow communication between members of the research team and the patient's outpatient clinician(s) (psychiatrist, psychotherapist, nurse practitioner, primary care physician, or equivalent) as needed to ensure safety
* Ability to safely participate in MRI
* Fluent in English

Exclusion Criteria:

* Imminent risk of suicide (based on the Columbia-Suicide Severity Rating Scale)
* Current depressive episode greater than or equal to 2 years duration
* Presence of primary psychiatric diagnoses other than MDD and/or comorbid generalized anxiety disorder (GAD) or phobia (e.g., post-traumatic stress disorder; obsessive-compulsive disorder; MDD w psychotic features; primary psychotic illness; Bipolar I or II)
* DSM-5 defined addiction to, dependence on, abuse of, or misuse of any substance during the prior 12 months, excluding nicotine
* Evidence of cognitive impairment (MMSE score falling greater than or equal to 1 SD below the mean score for his or her age and education)
* Recent onset (within 8 weeks of screening) psychotherapy, including, but not limited to: any form of treatment, aid, or therapy that has intensively and extensively examined the patient's psychological history, including, but not limited to: cognitive behavioral therapy, dialectical behavioral therapy, interpersonal therapy, and family-focused therapy
* Prior exposure to an adequate dose and duration of the TMS treatment protocol administered in this study during the current depressive episode.
* Participated in any clinical trial with an investigational drug or device within the past 6 weeks prior to screening
* History of neurosurgery to treat a neurological or psychiatric disorder
* Evidence or history of significant neurological disorder, including moderate-severe head trauma, stroke, Parkinson's disease or other movement disorder (except benign essential tremor), epilepsy, history of seizures, cerebrovascular disease, dementia, increased intracranial pressure, history of repetitive or severe head trauma, or primary or secondary tumors within the central nervous system
* Implanted electronic devices and/or conductive objects in or near the head, including metal plates, aneurysm coils, cochlear implants, ocular implants, deep brain stimulation devices and stents
* Any implanted device that is activated or controlled in any way by physiological signals, including, but not limited to: deep brain stimulators, cochlear implants, and vagus nerve stimulators
* Patients with major depressive disorder who have failed to receive clinical benefit from Vagus Nerve Stimulation (VNS) or are currently receiving these therapies.
* History of seizures (except juvenile febrile seizures) or any condition/concurrent medication that could notably lower seizure threshold
* Individuals who are pregnant, nursing, contemplating pregnancy within the length of the study or, in the opinion of the investigator, not adherent to a medically acceptable method of birth control
* History or presence of any disease, medical condition or physical condition that, in the opinion of the investigator, may compromise, interfere, limit, effect, or reduce the participant's ability to complete a treatment study lasting up to 21 weeks
* Abnormal bloodwork for electrolytes, thyroid and liver function
* Individuals who are taking > 300 mg daily dose of bupropion in any formulation (immediate, extended, or slow-release)
* Individuals who are taking tricyclic antidepressants.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in depression, as measured by the Hamilton Depression Rating Scale (HAMD17) | Baseline and 1 Week Post Treatment (8-10 weeks)
  The Hamilton Depression Rating Scale (HAMD17) is a 17 item clinician-rated measure of depression severity. Scores of 0-7 = Normal, 8-13 = Mild Depression, 14-18 = Moderate Depression, 19-22 = Severe Depression, ≥ 23 = Very Severe Depression

SECONDARY OUTCOMES:
Change in depression, as measured by the Quick Inventory of Depressive Symptomology (QIDS) | Baseline and Post Treatment (7-9 weeks)
  The Quick Inventory of Depressive Symptomology (QIDS) is a 16 item self-report measure of depression severity. Scores range from 0 to 27, with higher scores indicating greater severity of depression.
Change in Resting State fMRI Connectivity | Baseline and after completion of treatment (7-9 weeks)
  Calculated from Functional Magnetic Resonance Imaging (fMRI) scan conducted while participant is awake but not completing any tasks in the scanner. Used to determine biotype of depression for treatment assignment and to determine if any changes in resting state connectivity have taken place post-TMS treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Conor Liston, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
In accordance with NIH policy we will share our data via the National Database for Clinical Trials related to Mental Illness (NDCT). NDCT is a secure data platform that will allow us to share research data and tools from our analysis of resting-state fMRI data, task-based fMRI data, and fMRI-guided rTMS data. Specifically, data to be shared will include de-identified neuroimaging scans and rTMS targeting data, in addition to phenotypic data such as demographics, diagnosis, treatment history, and anonymized, item-level responses to clinical and cognitive assessments. These data will then be made available through the NDCT, and NIH-funded repository that ensures that data are secure and shared in accord with applicable NIH regulations.
Time Frame: Raw data (e.g., MRI data and assessment responses) will be deposited on the NDCT every six months (January 15 and June 15 of each year of the award period), in accordance with NIH policy for use of the NDCT in clinical trials research. Curated data will be uploaded annually beginning in the third year of the project.
Access Criteria: The data may be shared with researchers at institutions with a Federal Wide Assurance, who will be able to gain access to NDCT data by submitting a data access request, in line with NDCT policies.